CLINICAL TRIAL: NCT02869009
Title: Antiplatelet Therapy in Acute Mild-Moderate Ischemic Stroke (ATAMIS): a Parallel Randomized, Open-label, Multicenter, Prospective Study
Brief Title: Antiplatelet Therapy in Acute Mild-Moderate Ischemic Stroke
Acronym: ATAMIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of neurological department, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k2016-06
Record Dates: First submitted 2016-08-01; First posted 2016-08-16 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Ischemic Stroke
Keywords: stroke; clopidogrel; antiplatelets
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clopidogrel plus aspirin group (Experimental): the group will receive a 300mg loading dose of clopidogrel plus aspirin 100 mg, followed by clopidogrel 75 mg/d and aspirin 100 mg/d from day 2 to day 14, and followed by clopidogrel 75 mg/d or aspirin 100 mg/d from day 15 to day 90.
  Interventions: Drug: clopidogrel; Drug: Aspirin
- aspirin group (Experimental): the group will receive 100-300 mg aspirin from day 1 to day 14, followed by aspirin 100 mg/d from day 15 to day 90.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: clopidogrel
  Other Names: Plavix
  Arms: clopidogrel plus aspirin group
Drug: Aspirin

SUMMARY:
The risk of early recurrence or progression of acute ischemic stroke is very high, even in patients treated with aspirin. The Chance study show that clopidogrel plus aspirin treatment reduced the risk of recurrent stroke in patients with transient ischemic attack (TIA) or minor ischemic stroke (NIHSS ≤ 3) within 24 hour onset and was not associated with increased hemorrhage events, compared with aspirin monotherapy. However, it is not known whether the dual antiplatelet treatment could reduce the risk of early recurrence or progression in patients with acute mild to moderate ischemic stroke (4 ≤ NIHSS ≤ 10). The investigators hypothesise that clopidogrel-aspirin treatment will be superior to aspirin monotherapy in this group of patients.

DETAILED DESCRIPTION:
The ATAMIS study is a multicentre, prospective, randomised, open-label, controlled trial with a target enrollment of 3,000 patients from 60 centres of the Northeast China. Eligible patients are as follows: (1) definite acute ischemic stroke; (2) neurological deficit: 4 ≤ NIHSS ≤ 10; (3) time from onset to drug treatment: within 48 hours.

Patients in the clopidogrel-aspirin group will receive a 300mg loading dose of clopidogrel, followed by clopidogrel 75 mg/d and aspirin 75 mg/d from day 2 to day 14, and followed by clopidogrel 75 mg/d or aspirin 100 mg/d from day 15 to day 90.

Patients in the aspirin-alone group will receive 100-300 mg aspirin from day 1 to day 14, followed by aspirin 100 mg/d from day 15 to day 90.

The primary efficacy end point is early neurological deterioration assessed as a change of NIHSS: no change of NIHSS within 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Acute ischemic stroke that can be randomized within 48 hours of symptoms onset
* neurological deficit: 4 ≤ NIHSS ≤ 10
* CT or MRI scan ruling out hemorrhage or other pathology
* the first onset of ischemic stroke or previous stroke with no obvious sequelae (mRS≤1)
* Signed informed consent by patient self or legally authorized representatives

Exclusion Criteria:

* intracranial hemorrhage and hemorrhagic cerebral infarction
* Thrombolysis for ischemic stroke
* Allergy to clopidogrel and/or aspirin
* History of stroke with serious sequelae
* Severe systemic disease (such as severe infection, severe hepatic and renal dysfunction)
* Clear indication for anticoagulation (atrial fibrillation, mechanical cardiac valves, deep venous thrombosis, pulmonary embolism)
* History of intracranial hemorrhage
* Planned treatment with nonsteroidal anti-inflammatory drugs to affect platelet function
* Anticoagulation within 10 days
* Gastrointestinal bleed or major surgery within 3 months
* Planned or likely revascularization (any angioplasty or vascular surgery) within the next 3 months
* Planned surgery or intervention to stop antiplatelet therapy
* Ischemic stroke induced by angiography or surgery
* Pregnancy or childbirth within the previous 4 weeks
* Patients who have been treated with any other investigational drug within 3 months of enrollment
* Severe noncardiovascular comorbidity with life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Early neurological deterioration assessed as change of NIHSS | 14 days

SECONDARY OUTCOMES:
new clinical vascular events (ischemic stroke/hemorrhagic stroke/TIA/myocardial infarction/vascular death) | 90 days
Changes in National Institute of Health stroke scale scores | 14 days
moderate to severe bleeding events | 14 days
  cerebral hemorrhage，hemorrhage of digestive tract, or moderate to severe bleeding of other organs.
Total mortality | 90 days
Adverse events/severe adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Sheng Chen, Study Director — General Hospital of Shenyang Military Region; Xin-Hong Wang, Principal Investigator — General Hospital of Shenyang Military Region
Locations (1):
- General Hospital of Shenyang Military Region, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Wang Y, Zhao X, Liu L, Wang D, Wang C, Wang C, Li H, Meng X, Cui L, Jia J, Dong Q, Xu A, Zeng J, Li Y, Wang Z, Xia H, Johnston SC; CHANCE Investigators. Clopidogrel with aspirin in acute minor stroke or transient ischemic attack. N Engl J Med. 2013 Jul 4;369(1):11-9. doi: 10.1056/NEJMoa1215340. Epub 2013 Jun 26. PMID 23803136
- [Background] Wong KS, Chen C, Fu J, Chang HM, Suwanwela NC, Huang YN, Han Z, Tan KS, Ratanakorn D, Chollate P, Zhao Y, Koh A, Hao Q, Markus HS; CLAIR study investigators. Clopidogrel plus aspirin versus aspirin alone for reducing embolisation in patients with acute symptomatic cerebral or carotid artery stenosis (CLAIR study): a randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2010 May;9(5):489-97. doi: 10.1016/S1474-4422(10)70060-0. Epub 2010 Mar 22. PMID 20335070
- [Background] Kennedy J, Hill MD, Ryckborst KJ, Eliasziw M, Demchuk AM, Buchan AM; FASTER Investigators. Fast assessment of stroke and transient ischaemic attack to prevent early recurrence (FASTER): a randomised controlled pilot trial. Lancet Neurol. 2007 Nov;6(11):961-9. doi: 10.1016/S1474-4422(07)70250-8. Epub 2007 Oct 10. PMID 17931979
- [Background] Markus HS, Droste DW, Kaps M, Larrue V, Lees KR, Siebler M, Ringelstein EB. Dual antiplatelet therapy with clopidogrel and aspirin in symptomatic carotid stenosis evaluated using doppler embolic signal detection: the Clopidogrel and Aspirin for Reduction of Emboli in Symptomatic Carotid Stenosis (CARESS) trial. Circulation. 2005 May 3;111(17):2233-40. doi: 10.1161/01.CIR.0000163561.90680.1C. Epub 2005 Apr 25. PMID 15851601
- [Background] Bhatt DL, Fox KA, Hacke W, Berger PB, Black HR, Boden WE, Cacoub P, Cohen EA, Creager MA, Easton JD, Flather MD, Haffner SM, Hamm CW, Hankey GJ, Johnston SC, Mak KH, Mas JL, Montalescot G, Pearson TA, Steg PG, Steinhubl SR, Weber MA, Brennan DM, Fabry-Ribaudo L, Booth J, Topol EJ; CHARISMA Investigators. Clopidogrel and aspirin versus aspirin alone for the prevention of atherothrombotic events. N Engl J Med. 2006 Apr 20;354(16):1706-17. doi: 10.1056/NEJMoa060989. Epub 2006 Mar 12. PMID 16531616
- [Background] Diener HC, Bogousslavsky J, Brass LM, Cimminiello C, Csiba L, Kaste M, Leys D, Matias-Guiu J, Rupprecht HJ; MATCH investigators. Aspirin and clopidogrel compared with clopidogrel alone after recent ischaemic stroke or transient ischaemic attack in high-risk patients (MATCH): randomised, double-blind, placebo-controlled trial. Lancet. 2004 Jul 24-30;364(9431):331-7. doi: 10.1016/S0140-6736(04)16721-4. PMID 15276392
- [Derived] Yan HT, Cui Y, Li ZA, Cai JR, Wang Q, Hou XW, Chen HS. Effect of age on the efficacy and safety of clopidogrel plus aspirin vs aspirin alone in acute mild-to-moderate stroke: a secondary analysis of the ATAMIS trial. Front Neurol. 2025 Oct 27;16:1643517. doi: 10.3389/fneur.2025.1643517. eCollection 2025. PMID 41220961
- [Derived] Cui Y, Wang YH, Kong XR, Chen HS. Early Neurologic Deterioration and Efficacy of Dual Antiplatelet in Anterior Versus Posterior Circulation Stroke. J Am Heart Assoc. 2025 Feb 4;14(3):e037268. doi: 10.1161/JAHA.124.037268. Epub 2025 Jan 23. PMID 39846303
- [Derived] Cui Y, Liu QY, Chen HS. Dual Antiplatelet Therapy and Outcomes in Acute Mild to Moderate Stroke With Versus Without Large-Artery Atherosclerosis Post Hoc Analysis of ATAMIS. J Am Heart Assoc. 2024 Sep 17;13(18):e036318. doi: 10.1161/JAHA.124.036318. Epub 2024 Sep 9. PMID 39248249
- [Derived] Chen HS, Cui Y, Wang XH, Ma YT, Han J, Duan YJ, Lu J, Shen LY, Liang Y, Wang WZ, Wang H, Zhao Y, Zhang JT, Song YL, He XM, Li RH, Tao DB, Li J, Huang SM, Wang N, Hong M, Meng C, Zhang W, Wang DL, Nguyen TN; ATAMIS investigators. Clopidogrel Plus Aspirin vs Aspirin Alone in Patients With Acute Mild to Moderate Stroke: The ATAMIS Randomized Clinical Trial. JAMA Neurol. 2024 May 1;81(5):450-460. doi: 10.1001/jamaneurol.2024.0146. PMID 38466274
- [Derived] Hou X, Li X, Wang X, Chen H. Antiplatelet Therapy in Acute Mild-Moderate Ischemic Stroke (ATAMIS): a parallel, randomised, open-label, multicentre, prospective study. Stroke Vasc Neurol. 2018 Sep 23;3(4):263-267. doi: 10.1136/svn-2018-000148. eCollection 2018 Dec. PMID 30637134